CLINICAL TRIAL: NCT02708576
Title: A Phase 1 Randomized, Double Blind, Placebo Controlled, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of NGM313 in Healthy Overweight and Obese Adult Participants
Brief Title: Phase 1 Study of NGM313 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0201
Record Dates: First submitted 2016-02-29; First posted 2016-03-15 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NGM313 (Experimental): Administration of active NGM313
  Interventions: Biological: NGM313
- Placebo (Placebo Comparator): Administration of placebo comparator
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NGM313
  Arms: NGM313
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability of NGM313, both single dose and multiple doses, in normal healthy overweight and obese adult participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI range 27-40 kg/m2, inclusive for the SAD module, and 27-40 kg/m2, inclusive for the MAD module;
* Normal clinical laboratory evaluations
* Normal ECG findings

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* Uncontrolled hypertension defined as sitting blood pressure systolic > 150 mm/Hg and/or diastolic > 90 mm/Hg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Absolute change in weight in kilograms | 28 and 84 days

SECONDARY OUTCOMES:
Absolute change in fasting glucose in mmol/L | 28 and 84 days

OTHER OUTCOMES:
Safety and tolerability as measured by adverse events, vitals signs, electrocardiograms, and clinical laboratories | 28 and 84 days
Pharmacokinetics as measured by maximum observed concentration (cmax). | 28 and 84 days
Pharmacokinetics as measured by time to maximum concentration (tmax). | 28 and 84 days
Pharmacokinetics as measured by area under the curve (auc). | 28 and 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Que Liu, MD, Study Director — NGM Biopharmaceuticals, Inc
Locations (1):
- NGM Clinical Study Site, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No